CLINICAL TRIAL: NCT04865653
Title: LSD Base and LSD Tartrate Bioequivalence and Bioavailability in Healthy Subjects
Acronym: LSD-Bio
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2020-02331
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, 5-period cross-over design with five treatment conditions:
  1. Oral drinking solution of 0.1 mg LSD base in 96% ethanol
  2. Solid orodispersible film containing 0.1 mg LSD base
  3. Oral drinking solution of 0.146 mg LSD tartrate in water (equivalent to 0.1 mg LSD base)
  4. Intravenous administration of 0.146 mg LSD tartrate in water (equivalent to 0.1 mg LSD base)
  5. Placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Oral drinking solution of LSD base (Experimental): Oral drinking solution of 0.1 mg LSD base in 96% ethanol
  Interventions: Drug: Lysergic Acid Diethylamide Base oral drinking solution
- Solid orodispersible film containing LSD base (Experimental): Solid orodispersible film containing 0.1 mg LSD base
  Interventions: Drug: Lysergic Acid Diethylamide Base solid orodispersible film
- Oral drinking solution of LSD tartrate (Experimental): Oral drinking solution of 0.146 mg LSD tartrate in water
  Interventions: Drug: Lysergic Acid Diethylamide Tartrate oral drinking solution
- Intravenous administration of LSD tartrate (Experimental): Intravenous administration of 0.146 mg LSD tartrate in water
  Interventions: Drug: Lysergic Acid Diethylamide Tartrate intravenous administration
- Placebo (Placebo Comparator): Placebo for all formulations
  Interventions: Other: LSD Placebo

INTERVENTIONS:
Drug: Lysergic Acid Diethylamide Base oral drinking solution — A moderate dose of 0.1 mg LSD will be administered.
  Other Names: LSD
  Arms: Oral drinking solution of LSD base
Drug: Lysergic Acid Diethylamide Base solid orodispersible film — A moderate dose of 0.1 mg LSD will be administered.
  Other Names: LSD
  Arms: Solid orodispersible film containing LSD base
Drug: Lysergic Acid Diethylamide Tartrate oral drinking solution — A moderate dose of 0.146 mg LSD tartrate will be administered (equivalent to 0.1 mg LSD base).
  Other Names: LSD
  Arms: Oral drinking solution of LSD tartrate
Drug: Lysergic Acid Diethylamide Tartrate intravenous administration — A moderate dose of 0.146 mg LSD tartrate will be administered (equivalent to 0.1 mg LSD base).
  Other Names: LSD
  Arms: Intravenous administration of LSD tartrate
Other: LSD Placebo — Placebo for each formulation containing only the solvent or gel but no LSD.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Lysergic acid diethylamide (LSD) is used as recreational substance and as a research substance to study the mind. Recreationally, LSD is typically used in the form of "blotters" containing LSD tartrate. In research, both LSD base (LSD alone) or LSD salt in the form of LSD tartrate are used. The oral bioavailability of LSD is not known and LSD alone and LSD as salt have never been directly compared regarding their equivalence of plasma concentrations and effects. Because different forms of LSD are used in research it is important to know their difference or equivalence for correct dosing of LSD. The present study will compare equivalent doses of LSD base in ethanol orally, LSD tartrate in water administered orally, LSD base in an orodispersible film administered orally and LSD tartrate in water administered intravenously, as well as a placebo using a double-blind, randomized, counterballanced cross-over design in healthy participants.

DETAILED DESCRIPTION:
LSD is widely used for recreational and spiritual purposes. Additionally LSD is currently reused in experimental studies with healthy subjects and in studies investigating its effects on patients suffering from anxiety, depression, addiction personality disorders, cluster headache, migraine, and other pathological conditions.

When LSD is used recreationally, it is administered mostly in the form of LSD tartrate on filter paper (blotter) or as a liquid. In experimental research over the past years, LSD has mostly been used in the form of LSD base, which is lipophilic and therefore has typically been administered as a solution in ethanol. However, some researchers have also use LSD tartrate orally or LSD base intravenously. Currently, it is not clear how these different forms of LSD compare regarding their bioequivalence and effects.

The present study therefore compares four different formulations of LSD and placebo: (1) An oral drinking solution of LSD base currently used in many research studies (100 μg LSD in 96% ethanol), (2) A solid orodispersible film containing LSD base (100 μg LSD), (3) LSD tartrate used in research and recreationally (100 μg LSD equivalent of LSD tartrate in water), (4) an intravenous administration of LSD tartrate (100 μg LSD equivalent of LSD tartrate in water), and (5) placebo for all formulations (quadruple-dummy). The primary goals are to document the bioequivalence of LSD base (1) and tartrate (3) and to define the oral bioavailability of LSD using an additional intravenous LSD administration.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years old
2. Sufficient understanding of the German language
3. Understanding of procedures and risks associated with the study
4. Willing to adhere to the protocol and signing of the consent form
5. Willing to refrain from the consumption of illicit psychoactive substances during the study
6. Abstaining from xanthine-based liquids from the evenings prior to the study sessions to the end of the study days
7. Willing not to operate heavy machinery within 48 hours after substance administration
8. Willing to use double-barrier birth control throughout study participation
9. Body mass index between 18-29 kg/m2

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder
3. Psychotic disorder or bipolar disorder in first-degree relatives
4. Hypertension (>140/90 mmHg) or hypotension (SBP<85 mmHg)
5. Hallucinogenic substance use (not including cannabis) more than 20 times or any time within the previous two months
6. Pregnancy or current breastfeeding
7. Participation in another clinical trial (currently or within the last 30 days)
8. Use of medication that may interfere with the effects of the study medication
9. Tobacco smoking (>10 cigarettes/day)
10. Consumption of alcoholic beverages (>20 drinks/week)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
LSD plasma AUC | 18 months
  Assessed 22 times on each study day via blood samples
LSD Cmax | 18 months
  Assessed 22 times on each study day via blood samples
Bioavailability of LSD base | 18 months
  Assessed 22 times on each study day via blood samples
Bioavailability of LSD tartrate | 18 months
  Assessed 22 times on each study day via blood samples

SECONDARY OUTCOMES:
Acute subjective effects I | 18 months
  Visual Analog Scales (VAS) assessing the intensity and duration of subjective effects on a scale from 0% - 100% with higher scores representing more intense effects
Acute subjective effects II | 18 months
  5 Dimensions of Altered States of Consciousness (5D-ASC) consisting of 94 items to be rated on a visual analog scale (0-100 mm), with higher values indicating stronger effects
Acute subjective effects III | 18 months
  Spiritual Realm Questionnaire assesses the spiritual phenomenons elicited by psychedelic substances through 11 main questions to be answered on a total of 65 sub-ordered 100mm visual analog scales
Acute subjective effects IV | 18 months
  States of Consciousness Questionnaire assesses the emergence and intensity of phenomenons occurring in altered states of consciousness on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely")
Autonomic effects I | 18 months
  Assessed 23 times on each study day via systolic and diastolic blood pressure
Autonomic effects II | 18 months
  Assessed 23 times on each study day via heart rate
Autonomic effects III | 18 months
  Assessed 23 times on each study day via tympanic body temperature
Bioavailability of orodispersible film | 18 months
  Assessed 22 times on each study day via blood samples
NEO-Five-Factor-Inventory (NEO-FFI) | Baseline
  The NEO-FFI is a self-description questionnaire with 60 items for the measurement of the "big five": neuroticism, extraversion, openness, agreeableness, and consciousness. It uses a 5-point Likert scale ranging from "completely disagree" to "fully agree".
Freiburger Personality Inventory (FPI-R) | Baseline
  The FPI-R version comprises 138 items and covers 12 dimensions of personality: life satisfaction, social orientation, performance orientation, inhibition, excitability, aggressiveness, stress, physical complaints, health concerns, openness, as well as the secondary factors according to Eysenck's Extraversion and Emotionality (Neuroticism). It uses a 2-point scale ("true" and "not true").
Saarbrücker Personality Questionnaire (SPF) | Baseline
  The SPF defines empathy as the "reactions of one individual to the observed experiences of another." It assesses 28-items on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well". The measure has 4 subscales (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) each made up of 7 different items.
HEXACO personality inventory | Baseline
  The HEXACO personality inventory is a six-dimensional model of human personality with 100 items.The six factors are: Honesty-Humility, Emotionality, Extraversion, Agreeableness, Conscientiousness and Openness to Experience. The HEXACO uses a 5-point Likert scale ranging from "completely disagree" to "fully agree".
Defense Style Questionnaire (DSQ-40) | Baseline
  The DSQ-40 can provide scores for 20 individual defenses, and scores for the three factors "mature", "neurotic", and "immature". Each item is evaluated on a scale from 1 to 9, where "1" indicates "completely disagree" and "9" indicates "fully agree".
Absence of tolerance | 18 months
  Absence of tolerance (no significant order effect) with repeated dosing of LSD with a between dosing interval of at least 10 days assessed with Visual Analog Scales (any drug response over time)
Appreciation Scale (AS) | Baseline
  The Appreciation Scale comprises 57 items used to measure eight aspects of appreciation. The eight subscales are respectively focus on what one has ("Have" Focus), Awe, Ritual, Present Moment, Self/Social Comparison, Gratitude, Loss/Adversity, and Interpersonal. Each item is evaluated on a scale from 1 to 7 in terms of either attitude intensity ("strongly disagree" to "strongly agree") or frequency ("never" to "more than once a day").
Subjective well-being I | 18 months
  The Scale of Positive and Negative Experience (SPANE) is a 12-item questionnaire to capture the affective component of subjective well-being. It includes six items to assess positive feelings and six items to assess negative feelings. The feelings are reported on a 5-point scale ranging from "very rarely" to "very often or always".
Subjective well-being II | 18 months
  The Positive Attitude towards life is an 8-item subscale of the 39-item Bern Subjective Well-Being Questionnaire and assesses different dimensions of subjective well-being. Evaluations are made using a six-point rating scale ranging from 1 ("strongly disagree") to 6 ("strongly agree").
Subjective well-being III | 18 months
  Global Life Satisfaction (GLS) is assessed on a single item life satisfaction measure. The question is answered on a 11-point scale with 0 as "not at all satisfied with your life" and 10 " completely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Clinical Pharmacology & Toxicology, University Hospital Basel, Basel, Switzerland